CLINICAL TRIAL: NCT04727203
Title: Active and Healthy Ageing for All: a Multi-component Healthy Lifestyle Program (AHAA)
Brief Title: Active and Healthy Ageing for All: a Multi-component Healthy Lifestyle Program
Acronym: AHAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Odisee University college for applied sciences (Other)
Responsible Party: Principal Investigator, Julie Vanderlinden, Phdc, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AHAA
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Health Promotion
Keywords: ageing; healthy lifestyle; intervention
MeSH Terms: interventions — Exercise; Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Intervention Model Description: There are 6 groups in this intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Partcipants in this group will receive the 8 week healthy lifestyle program
  Interventions: Behavioral: AHAA
- Control (No Intervention): Participants in this group will not receive any intervention

INTERVENTIONS:
Behavioral: AHAA — Multi-component healthy lifestyle program
  Other Names: Active and healthy ageing for all
  Arms: Intervention

SUMMARY:
AHAA is a healthy lifestyle program offered to older adults aged 60+ years. The program is developed based upon co-creation with the target group and implemented and evaluated in several locations.

DETAILED DESCRIPTION:
1. co-creation : all participants will be questioned and included in the co-creation session
2. implementation : the developed multicomponent healthy lifestyle program will be enrolled and implemented in 6 locations (community services for older adults in Flanders and Brussels)
3. evaluation : the program will be evaluated (effects and process)

ELIGIBILITY:
Inclusion Criteria:

* age 60+ years

Exclusion Criteria:

* not being able to attend the weekly meetings

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity measured by IPAQ | up to twelve weeks
  Subjective physical activity
Physical activity measured by accelerometry | up to twelve weeks
  Objective physical activity
Sedentary behaviour measured by accelerometry | up to twelve weeks
  Objective sedentary behaviour
Sedentary behaviour measured by IPAQ | up to twelve weeks
  Subjective sedentary behaviour
Nutrition questionnaire (self-reported) | up to twelve weeks
  Nutrition
Sleep measured by accelerometry | up to twelve weeks
  Objective sleep
Sleep measured by PSQI | up to twelve weeks
  Subjective sleep

SECONDARY OUTCOMES:
well-being measured by WEMWBS | up to twelve weeks
  well-being
Perceived stress measured by the perceived stress scale | up to twelve weeks
  Perceived stress of participants
Perceived positive health status measured by a self-reported questionnaire | up to twelve weeks
  Perceived positive health status
Health literacy measured by HLSQ self-reported questionnaire | up to twelve weeks
  Health literacy
Social support measured by a self-reported questionnaire | up to twelve weeks
  Social Support

CONTACTS AND LOCATIONS:
Overall Officials: Julie Vanderlinden, PHDc, Principal Investigator — KU Leuven
Locations (5):
- Belgium (5):
  - LDC, Aalst
  - LDC, Brussels
  - Regie Ouderenzorg, Ghent
  - LDC, Mechelen
  - Triamant, Sint-Truiden

IPD SHARING:
Plan to Share IPD: No